CLINICAL TRIAL: NCT06947837
Title: Study on the Influencing Mechanism and Promoting Strategies of Post-partum Nurses' Work Engagement
Acronym: Nurses
Status: Completed | Type: Observational
Sponsor: keqin liu (Other)
Responsible Party: Sponsor-Investigator, keqin liu, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202503043; 2024C06 (Other: Tongji Hospital affiliated to Huazhong University of Science and Technology)
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Nurses; Postpartum; Work Engagement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of postpartum returning nurses: The cohort of postpartum returning nurses mainly included nurses who worked in clinical practice after maternity leave and voluntarily participated in this study. The study time was 1 month, 3 months and 6 months after postpartum return to work, and mainly included basic information, social support, postpartum return to work, sleep and psychological status follow-up survey.

SUMMARY:
The goal of this observational study is to through the combination of longitudinal qualitative research and longitudinal quantitative research, the work experience changes of nurses returning to work after delivery were analyzed, and the changing trajectory and influencing mechanism of work involvement of nurses returning to work after delivery were explored.On this basis, combined with the existing literature, the promotion strategy of post-natal nurses' work involvement was constructed in order to improve the level of post-natal nurses' work involvement, help them better adapt to clinical nursing work, and improve the quality of nursing service.

ELIGIBILITY:
Inclusion Criteria:

* Nurses returning to work after childbirth are engaged in clinical nursing work in the hospital;
* The time to return to work after childbirth is less than 1 month;
* Informed and voluntary participation in the study.

Exclusion Criteria:

* Training, rotation, practice nurses;
* Give birth to abnormal children.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nurses from Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology who returned to work within 1 month after delivery were selected.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-09-30 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Postpartum work engagement | Through study completion, an average of 1 year (the specific follow-up time was 1 month, 3 months and 6 months after delivery).
  We used "Utreeht Work Engagement Scale" to measure and evaluate the work engagement of postpartum nurses return to work. The Work Engagement Scale indicated the higher the score, the greater the work engagement.

SECONDARY OUTCOMES:
Social Support situation | Through study completion, an average of 1 year (the specific follow-up time was 1 month, 3 months and 6 months after delivery).
  We used "Development and psychometric properties of a perceived social support scale for nurses returning to work after childbirth" to evaluate the social support of postpartum returning nurses. The scale showed that the higher the score, the greater the social support.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Liu, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No